CLINICAL TRIAL: NCT04499937
Title: ReCoUPS: Incentive-Based and Real-Time Symptom and Activity Reporting After Concussion
Brief Title: ReCoUPS: Post-Concussion Patient Reports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-013326
Record Dates: First submitted 2020-07-20; First posted 2020-08-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Brain Concussion; Head Injury
MeSH Terms: conditions — Brain Concussion; Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Streak incentive (Experimental): Subjects start with no money in an account, but they earn a fixed amount with each response. In this arm, each adult report is worth $3.17 so an adult subject can earn up to $200 if he/she responds to all surveys. If an adult completes at least 75% of the reports, he/she will receive an $100 bonus for a total maximum of $300. In this arm, each child report is worth 0.52 cents so a child subject can earn up to $33 if he/she responds to all surveys. If a child completes at least 75% of the reports, he/she will receive a $17 bonus for a total maximum of $50.
  Interventions: Behavioral: Streak incentive
- Loss-based incentive (Experimental): Subjects start with the maximum possible compensation, but money is deducted for each missed response. Adult subjects will lose $4.76 for each missed survey. Child subjects will lose $0.79 for each missed survey.
  Interventions: Behavioral: Loss-based incentive
- Flat-fee control status quo condition (Active Comparator): Subjects will receive the maximum possible compensation at the end of the study regardless of response rate.
  Interventions: Behavioral: Flat-fee control status quo condition
- Flat-Fitbit control status quo condition (Active Comparator): Subjects will be compensated by keeping the Fitbit at the end of the study regardless of response rate.
  Interventions: Behavioral: Flat-Fitbit control status quo condition

INTERVENTIONS:
Behavioral: Streak incentive — Participants will receive prompts 3 times a day for 21 days prompting them to complete surveys. They will start with a $0 balance and will earn a fixed amount for each response.
  Arms: Streak incentive
Behavioral: Loss-based incentive — Participants will receive prompts 3 times a day for 21 days prompting them to complete surveys. They will start with the maximum balance and will lose a fixed amount for each response they do not complete.
  Arms: Loss-based incentive
Behavioral: Flat-fee control status quo condition — Participants will receive prompts 3 times a day for 21 days prompting them to complete surveys. They will receive the maximum compensation at the end of the study.
  Arms: Flat-fee control status quo condition
Behavioral: Flat-Fitbit control status quo condition — Participants will receive prompts 3 times a day for 21 days prompting them to complete surveys. They will keep the Fitbit at the end of the study.
  Arms: Flat-Fitbit control status quo condition

SUMMARY:
Physical and cognitive rest are recommended as treatment for concussion, but debate persists about the utility of this recommendation for patients recovering from concussion. In addition, patient adherence to physical and cognitive rest recommendations after concussion remains unknown. This study will measure and compare symptom and activity reports in the days and weeks after a concussion among patients randomly assigned to different incentive-based arms.

DETAILED DESCRIPTION:
Although physical and cognitive rest are recommended as the hallmark treatment for concussion, debate persists about the utility of this recommendation for patients recovering from a concussion. In addition, patient adherence to physical and cognitive rest recommendations after concussion remains unknown. Objective and timely measures of physical and cognitive activity will aid in defining the relationship between physical and cognitive rest and clinical outcomes, such as symptom status, in the days and weeks after a concussion. Random assignment to incentive-based arms will be used to measure patient engagement with the study protocol and a dedicated research platform that involves ecological momentary assessment (EMA), in which participants report their real-time symptoms and daily activities in response to randomly timed prompts, will be used to help assess the rest and recovery process among pediatric and adult patients after concussion.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 13 to 64 years.
* Presents with head injury concerning for concussion in line with criteria specified in the most recent Consensus Statement on Concussion in Sport, defined as head trauma with neurologic impairment, including, but not limited to somatic (eg, headache), cognitive (eg, feeling like in a fog) and/or emotional symptoms (eg, lability) symptoms.
* Within approximately 5 days of injury.
* Ownership of a smartphone to report symptoms and activities.
* Speak English.
* Informed consent or parental/guardian permission and child assent for those under 18 years of age.

Exclusion Criteria:

* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 13 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Participant adherence to completing daily survey | 21 days
  This is a study where each participant is sent a short survey (PCSI instrument) three times each day for 21 days. The participant is instructed to reply to each survey within several minutes of receiving the prompt. We are interested in the extent to which participants will adhere to this instruction. Therefore, the outcome of interest is whether or not the participant replied to a given survey prompt. When we evaluate patient adherence in the data, we do this by calculating the % of survey prompts to which a given participant responded. In sum, the outcome is adherence to the survey.

SECONDARY OUTCOMES:
Time to recovery | 1 to 21 days
  Assess and quantify the concussion recovery process by monitoring symptoms and cognitive and physical activity on a daily basis.
Correlation between symptoms and physical activity | 1-21 days
  Determine if there is a correlation each day between the daily symptom score from the PCSI (0-126) and the number of hours spent exercising (physical activity).
Patient-reported activity vs. objective measures of activity | 1-21 days
  Compare the patient-reported hours spent exercising on a given day to the patient's daily step count collected through Fitbit on that same day.
Test Way to Health platform | 1-21 days
  Test Way to Health as a platform for efficiently randomizing and monitoring patients
Correlation between symptoms and cognitive activity | 1-21 days
  Determine if there is a correlation each day between the daily symptom score from the PCSI (0-126) and the number of hours participants spent doing homework, napping, and using screens combined (cognitive activity).

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Wiebe, PhD, Principal Investigator — University of Pennsylvania; Daniel Corwin, MD, Principal Investigator — Children's Hospital of Philadelphia; Christina Master, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korley FK, Kelen GD, Jones CM, Diaz-Arrastia R. Emergency Department Evaluation of Traumatic Brain Injury in the United States, 2009-2010. J Head Trauma Rehabil. 2016 Nov/Dec;31(6):379-387. doi: 10.1097/HTR.0000000000000187. PMID 26360006
- [Background] McCrea M, Guskiewicz KM, Marshall SW, Barr W, Randolph C, Cantu RC, Onate JA, Yang J, Kelly JP. Acute effects and recovery time following concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2556-63. doi: 10.1001/jama.290.19.2556. PMID 14625332
- [Background] Leddy JJ, Baker JG, Kozlowski K, Bisson L, Willer B. Reliability of a graded exercise test for assessing recovery from concussion. Clin J Sport Med. 2011 Mar;21(2):89-94. doi: 10.1097/JSM.0b013e3181fdc721. PMID 21358497
- [Background] Brown NJ, Mannix RC, O'Brien MJ, Gostine D, Collins MW, Meehan WP 3rd. Effect of cognitive activity level on duration of post-concussion symptoms. Pediatrics. 2014 Feb;133(2):e299-304. doi: 10.1542/peds.2013-2125. Epub 2014 Jan 6. PMID 24394679
- [Background] McCrory P, Meeuwisse WH, Aubry M, Cantu B, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen RG, Guskiewicz K, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport: the 4th International Conference on Concussion in Sport held in Zurich, November 2012. Br J Sports Med. 2013 Apr;47(5):250-8. doi: 10.1136/bjsports-2013-092313. No abstract available. PMID 23479479
- [Background] Moor HM, Eisenhauer RC, Killian KD, Proudfoot N, Henriques AA, Congeni JA, Reneker JC. The relationship between adherence behaviors and recovery time in adolescents after a sports-related concussion: an observational study. Int J Sports Phys Ther. 2015 Apr;10(2):225-33. PMID 25883871
- [Background] Meehan WP 3rd, Bachur RG. The recommendation for rest following acute concussion. Pediatrics. 2015 Feb;135(2):362-3. doi: 10.1542/peds.2014-3665. Epub 2015 Jan 5. No abstract available. PMID 25560439
- [Background] Thomas DG, Apps JN, Hoffmann RG, McCrea M, Hammeke T. Benefits of strict rest after acute concussion: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):213-23. doi: 10.1542/peds.2014-0966. Epub 2015 Jan 5. PMID 25560444
- [Background] Schneider KJ, Iverson GL, Emery CA, McCrory P, Herring SA, Meeuwisse WH. The effects of rest and treatment following sport-related concussion: a systematic review of the literature. Br J Sports Med. 2013 Apr;47(5):304-7. doi: 10.1136/bjsports-2013-092190. PMID 23479489
- [Background] Wiebe DJ, Nance ML, Houseknecht E, Grady MF, Otto N, Sandsmark DK, Master CL. Ecologic Momentary Assessment to Accomplish Real-Time Capture of Symptom Progression and the Physical and Cognitive Activities of Patients Daily Following Concussion. JAMA Pediatr. 2016 Nov 1;170(11):1108-1110. doi: 10.1001/jamapediatrics.2016.1979. No abstract available. PMID 27617669
- [Derived] Corwin DJ, Orchinik J, D'Alonzo B, Agarwal AK, Pettijohn KW, Master CL, Wiebe DJ. A Randomized Trial of Incentivization to Maximize Retention for Real-Time Symptom and Activity Monitoring Using Ecological Momentary Assessment in Pediatric Concussion. Pediatr Emerg Care. 2023 Jul 1;39(7):488-494. doi: 10.1097/PEC.0000000000002870. Epub 2022 Nov 3. PMID 36730797